CLINICAL TRIAL: NCT01174303
Title: A Trial Investigating the Pharmacodynamic Properties of NN5401 in Young Adults and Geriatric Subjects With Type 1 Diabetes
Brief Title: A Trial Investigating the Exposure of NN5401 in Young Adults and Elderly Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-1981; U1111-1114-9373 (Other: WHO); 2009-017280-42 (EudraCT Number)
Record Dates: First submitted 2010-08-02; First posted 2010-08-03 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec, insulin aspart drug combination; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp - BIAsp (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart; Drug: biphasic insulin aspart 30
- BIAsp - IDegAsp (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart; Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Each subject will be randomly allocated to two single doses injected subcutaneously (under the skin) of insulin degludec/insulin aspart and biphasic insulin aspart 30 in random order.
Drug: biphasic insulin aspart 30 — Each subject will be randomly allocated to two single doses injected subcutaneously (under the skin) of insulin degludec/insulin aspart and biphasic insulin aspart 30 in random order.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the exposure of NN5401 (insulin degludec/insulin aspart) in young adults and elderly subjects with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-35 years (both inclusive) (young group) or at least 65 years (geriatric group)
* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.0-28.0 kg/m^2 (both inclusive)
* HbA1c (glycosylated haemoglobin A1c) maximum 10.0% by central laboratory analysis

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Area under the Glucose Infusion Rate curve (only for NN5401) | from 0 to 24 hours after single-dose administration

SECONDARY OUTCOMES:
Area under the glucose infusion rate curve (only for biphasic insulin aspart 30) | from 0 to 24 hours after single-dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- [Result] Brunner M, Pieber T, Korsatko S, Kojzar H, Svendsen AL, Haahr H. The Distinct Prandial and Basal Pharmacodynamics of IDegAsp Observed in Younger Adults Are Preserved in Elderly Subjects with Type 1 Diabetes. Drugs Aging. 2015 Jul;32(7):583-90. doi: 10.1007/s40266-015-0272-y. PMID 26088815
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com